CLINICAL TRIAL: NCT07381413
Title: Eye Tracking Study on Eye Movement Function and Visual Attention Patterns in Patients With Thyroid-Associated Ophthalmopathy
Acronym: TAO-A
Status: Recruiting | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Ruili Wei, Chief of Ophthalmology, Shanghai Changzheng Hospital
Other Study IDs: TAO-A
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Thyroid Associated Ophthalmopathies; Eye Tracking
Keywords: TAO; eye tracking
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAO
  Interventions: Device: Non-invasive Eye Tracking Assessment
- CON
  Interventions: Device: Non-invasive Eye Tracking Assessment

INTERVENTIONS:
Device: Non-invasive Eye Tracking Assessment — This is an observational study; no therapeutic intervention is administered. All participants undergo a single, standardized study visit that includes:
  Participants will undergo a visual function assessment using a desktop-based high-frequency eye tracker. The assessment consists of three parts:
  1. Calibration: To ensure accurate gaze tracking.
  2. Oculomotor Tasks: Participants track visual targets to measure fixation stability and smooth pursuit capabilities.
  3. Visual Attention Tasks: Participants view static images to record scanning patterns.
  The entire process is non-invasive and lasts approximately 15-20 minutes.

SUMMARY:
This study focuses on eye health and visual function in patients with Thyroid-Associated Ophthalmopathy (TAO), a condition that often causes bulging eyes and restricted eye movement. The purpose of this study is to use non-invasive eye-tracking technology to evaluate how the disease affects eye movement function. The investigators hypothesize that compared to healthy individuals, patients with TAO will show measurable differences in eye stability and the ability to track moving objects. Additionally, the investigators believe the disease may alter how patients visually scan faces (e.g., avoiding eye contact). The study will enroll 100 participants, including both patients and healthy volunteers. By recording gaze patterns while participants look at a screen, the investigators aim to objectively quantify the physical and social impact of the disease, providing better data for future treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years, inclusive.
* Willing and able to provide written informed consent.
* Best-corrected visual acuity (BCVA) ≥ 1.0 in both eyes, with no history of ocular diseases or thyroid disorders.

Exclusion Criteria:

* Non-TAO Ocular Motility Disorders: History of conditions like myasthenia gravis, cranial nerve palsy, or congenital strabismus.
* Neurological Diseases: Disorders affecting oculomotor control (e.g., Parkinson's, MS, stroke, or brain tumors).
* Significant Visual Impairment: BCVA < 0.5 due to media opacities or retinopathy, preventing clear visualization of stimuli.
* Prior Ocular Surgery: History of surgeries affecting extraocular muscle mechanics (e.g., strabismus surgery, scleral buckling).
* Psychiatric or Cognitive Disorders: Inability to follow instructions or conditions affecting eye movements (e.g., schizophrenia).
* Medication Interference: Use of drugs affecting reaction time (e.g., sedatives) within 48 hours of testing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Thyroid-Associated Ophthalmopathy (TAO) group will consist of consecutive patients presenting to the clinic who are diagnosed with TAO according to the 2022 Chinese Guidelines for the Diagnosis and Treatment of Thyroid-Associated Ophthalmopathy. The healthy control group will be recruited through hospital staff volunteers and community advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-31 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Smooth Pursuit Function Gaze Distribution | Baseline
  Participants track a moving target on the screen. This metric quantifies the spatial distribution of fixation points recorded throughout the task duration

SECONDARY OUTCOMES:
Central Fixation Stability | Baseline
  This outcome measures the participant's ability to maintain a steady gaze on a central target for a predefined duration. It is quantified by the percentage of fixation time remaining within a small predefined area around the target center.
Gaze Distribution on Ocular Areas of Interest | Baseline
  This metric analyzes the visual attention patterns when viewing images.This is used to evaluate potential social-visual avoidance or altered scanning strategies in TAO patients compared to healthy controls.
Extraocular Muscle (EOM) Thickness | Baseline
  The thickness of the extraocular muscles (including the medial, lateral, superior, and inferior rectus). This anatomical metric serves as a biological marker of disease severity and will be correlated with eye-tracking functional data to explore the relationship between muscle hypertrophy and movement impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Changzheng Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No